CLINICAL TRIAL: NCT07073703
Title: Effectiveness of a Personalized 6-month Programme on Frailty in Older Patients Treated for Bladder or Kidney Cancer - FRAGECO - Multicenter, Controlled, Randomized Study
Brief Title: Effectiveness of a Personalized 6-month Programme on Frailty in Older Patients Treated for Bladder or Kidney Cancer.
Acronym: FRAGECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24CH124; 2024-A01991-46 (Other: ANSM)
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Kidney (Renal Cell) Cancer
Keywords: Exercise; Older people; Cancer; Bladder; Kidney; Frailty; Surgery
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell; Motor Activity; Frailty | interventions — diacetamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will consist of patients with bladder or kidney cancer receiving standard care, which includes a comprehensive assessment by an oncogeriatrician followed by surgery approximately 4 weeks later. Postoperatively, patients will be transferred to a rehabilitation center (SSR) for recovery, in line with standard clinical practice.
  As part of the study protocol, control group patients will undergo additional follow-up assessments alongside their usual care. These follow-ups-conducted at baseline, and at 1, 2, 3 months, and at the final endpoint-will mirror those of the intervention group. They will include patients- completed questionnaires and physical assessments conducted by an adapted physical activity teacher.
- Interventional group (Experimental): The interventional group will consist of bladder and kidney cancer patients who will follow a personalized 6-month care pathway in addition to standard care. This pathway includes:
  * 2 adapted physical activity (APA) sessions per week for 4 weeks prior to surgery
  * 2 APA sessions/ week for 4 weeks following surgery
  * Therapeutic education workshops tailored to individual needs, covering topics as physical activity, nutrition, treatments, fatigue, and relaxation
  * Referral to the department's DAPAP for a 12-week "bridge program", consisting of one APA session per week.
  The study will be conducted in the oncogeriatrics departments of Saint-Etienne University Hospital and Loire Private Hospital.
  Interventions: Procedure: APA; Behavioral: Therapeutic education workshops; Procedure: DAPAP

INTERVENTIONS:
Procedure: APA — 2 adapted physical activity (APA) sessions per week for 4 weeks before and after surgery
  Arms: Interventional group
Behavioral: Therapeutic education workshops — Therapeutic education workshops tailored to individual needs, covering topics as physical activity, nutrition, treatments, fatigue, and relaxation.
  Arms: Interventional group
Procedure: DAPAP — Referral to the department's DAPAP for a 12-week "bridge program", consisting of one session per week.
  Arms: Interventional group

SUMMARY:
Bladder and kidney cancers are commonly diagnosed in older adults. Surgery remains the primary treatment modality for patients with kidney or bladder cancer. In older patients, common co-morbidities include fatigue, physical deconditioning characterized by reduced cardiorespiratory fitness and progressing sarcopenia, pain- whether disease- related or treatment-induced- and undernutrition. These factors increased the risk of post-operative complications and exacerbate patient frailty.

The investigators propose a personalized 6-month program both pre- and post-surgery, including adapted physical activity sessions, therapeutic education workshops, and systematic referral to the department's DAPAP program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bladder or kidney cancer
* Surgical treatment
* No severe cognitive impairment preventing understanding of the protocol
* Affiliated or entitled to a social security scheme
* Having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Surgery already done
* Significant co-morbidities that contraindicate physical activity: associated cardiac pathologies, respiratory pathologies, disabling joint pathologies, etc.
* Deprived of liberty or under guardianship
* Benefiting from a prehabilitation prescription with a private physiotherapist.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Patient frailty | Day : 1 and Month : 6
  Frailty will be measured using the walking distance (in metres) achieved during the 6-minute walk test (6MWT) 6 months after the patient's inclusion.

SECONDARY OUTCOMES:
Cumulative Illness Rating Scale for Geriatrics (CIRS-G) | Months : 1, 2, 3 and 6
  The CIRS (Cumulative Illness Rating Scale) score provides a relevant comparison of the medical burden and treatment outcomes in geriatric patients with variable and complex pathologies.
  The score ranges from 0: no problem to 4: very serious problem.
Fried's frailty phenotype (FP) | Months : 1, 2, 3 and 6
  Frailty will be measured using Fried's frailty phenotype (FP), defined by exhaustion (EX), unexplained weight loss (WL), weakness (WK), sluggishness (SL) and low physical activity (LA). Three or more components define the frailty state, and one or two the pre-fragility state.
level of physical activity | Months : 1, 2, 3 and 6
  Objective measures of PA (in MET-hours/week) via accelerometry (Actigraph GT3x, Pensacola, Florida, USA) and subjective measurements of PA (in METhours/week) using the e-Adult Physical Activity Questionnaire (EA SNA-EPIS, Université Jean Monnet, Saint-Etienne, France).
level of sedentary lifestyle | Months : 1, 2, 3 and 6
  Objective measures of sedentary time (in h/d) via accelerometry (Actigraph GT3x, Pensacola, Florida, USA) and subjective measurements of sedentary behaviour (in hours/day) using the e-Adult Physical Activity Questionnaire (EA SNA-EPIS, Université Jean Monnet, Saint-Etienne, France).
Nutritional status | Months : 1, 2, 3 and 6
  With the Mini Nutritional Assessment (MNA) and albumin analysis in g/l, a level <35g/l: undernutrition, <30g/l: severe undernutrition.
Memory | Months : 1, 2, 3 and 6
  Mini-Mental State Examination (MMSE), which consists of 30 questions and is scored out of 30. The severity of memory impairment is considered mild if the score is above 20, moderate if the score is between 10 and 20, and severe if the score is below 10.
Healthy quality of life | Months : 1, 2, 3 and 6
  With the EORTC-QLC30 version 3. This 30-item questionnaire assesses 15 dimensions of quality of life (5 functional scales: physical, cognitive, social, emotional or psychological and limitations in daily activities; 1 global health/quality of life scale; 9 symptom scales: fatigue, nausea and vomiting, pain, dyspnea, insomnia, loss of appetite, constipation and diarrhea, financial problems related to the disease).
Fatigue | Months : 1, 2, 3 and 6
  With the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F). The questionnaire consists of 13 questions, each of which corresponds to a Likert scale ranging from 0 to 4 (0 = not at all, 4 = very much). A score is obtained out of 52, with the higher the score, the less fatigued the patient is.
Depression | Months : 1, 2, 3 and 6
  Using the Mini Geriatric Depression Scale (GDS) to 4 questions. If the score is greater than 1: high probability of depression, if the score is 0: high probability of no depression.
Muscular strength | Months : 1, 2, 3 and 6
  Muscle strength (in kilogram) on the handgrip.
Balance | Months : 1, 2, 3 and 6
  Assessed using the time (in seconds) taken to complete the Timed Up and Go (TUG). A time ≥ 20 seconds is associated with a risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU de Saint Etienne
Locations (2):
- France (2):
  - Chu Saint-Etienne, Saint-Etienne
  - Hôpital privé de la Loire, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No